CLINICAL TRIAL: NCT01223677
Title: Randomized Controlled Trial Evaluating Two Versions of a Rumination-focused CBT Training for the Presence of Depression and Anxiety in Adolescents and Young Adults
Brief Title: Rumination-focused CBT Training for the Prevention of Depression and Anxiety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Thomas Ehring, PhD., Universität Münster
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 50-50105-96-635
Record Dates: First submitted 2010-10-12; First posted 2010-10-19 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Depression; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rumination focused CBT (Active Comparator): RFCBT-group. This group training is based on research showing that dysfunctional forms of rumination are characterized by an abstract evaluative style of processing, whereas functional forms of of processing are more concrete and process-focused. The training uses psycho-education, functional analysis, group discussion, experiential exercises and behavioral experiments to facilitate the shift from dysfunctional ruminative thinking to a more helpful concrete thinking style.
  Interventions: Behavioral: Rumination Focused CBT
- rumination focused CBT (online) (Active Comparator): The online training is based on research showing that dysfunctional forms of rumination are characterized by an abstract evaluative style of processing, whereas functional forms of of processing are more concrete and process-focused. The training uses psycho-education, functional analysis, experiential exercises and behavioral experiments to facilitate the shift from dysfunctional ruminative thinking to a more helpful concrete thinking style.
  Interventions: Behavioral: Rumination Focused CBT
- No training control group (No Intervention): No training control group. Participants within this condition received no treatment, but only filled out the outcome measures at each measurement period.

INTERVENTIONS:
Behavioral: Rumination Focused CBT — see arms
  Other Names: RFCBT
  Arms: rumination focused CBT; rumination focused CBT (online)

SUMMARY:
Depression and anxiety disorders are highly prevalent and associated with reduced quality of life for patients and enormous economic costs for society. Although effective treatments are available, a substantial number of patients fail to respond, and the time between disorder onset and treatment is typically long. The development of prevention programs therefore appears promising. The current project aims to prevent depression and anxiety by targeting excessive levels of worry and rumination, two important risk factors for emotional disorders. Participants will be selected on the basis of a high score on two validated questionnaires on worry and rumination. They will be randomly assigned to a rumination-focused cognitive-behavioral training delivered in a group format, a rumination-focused cognitive-behavioral training delivered via internet, or a no-training control condition. It is expected that both versions of the rumination-focused training will reduce symptoms of depression and anxiety, will reduce the incidence of major depressive episodes and generalized anxiety disorder, and will reduce symptom levels of other emotional disorders.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* A score above the 75% and 66.7% percentile on two validated self-report measures of rumination and worry, the Ruminative Response Scale of the Response Style Questionnaire (RSQ; Nolen-Hoeksema & Morrow, 1991), and the Penn State Worry Questionnaire (PSWQ; Meyer et al. 1990).

Exclusion Criteria:

* A score indicating fulfillment of DSM-IV criteria for depression or generalized anxiety disorder according to the Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001) or the Generalized Anxiety Disorder Questionnaire-IV (GADQ-IV; Newman et al., 2002)

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 251 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory II (BDI-II) | 1 year after training has ended
  self-report questionnaire of depressive symptom severity

SECONDARY OUTCOMES:
Mood and Anxiety Symptom Questionnaire (MASQ-30) | 1 year after training has ended
  Symptom severity of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ehring, PhD, Principal Investigator — Westfalische Wilhelms Universitat Munster
Locations (1):
- University of Amsterdam, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Watkins ER, Moberly NJ. Concreteness training reduces dysphoria: a pilot proof-of-principle study. Behav Res Ther. 2009 Jan;47(1):48-53. doi: 10.1016/j.brat.2008.10.014. Epub 2008 Oct 21. PMID 19036353